CLINICAL TRIAL: NCT03435068
Title: The Evaluation of Soft Tissue Wound Healing Following Different Gingivectomy Applications: A Prospective Randomized Clinical Trial
Brief Title: Soft Tissue Wound Healing Following Different Gingivectomy Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: T.C. Dumlupınar Üniversitesi (Other)
Responsible Party: Principal Investigator, Berceste Guler, Assist .Prof, T.C. Dumlupınar Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-KAEK-86/05-39
Record Dates: First submitted 2018-02-04; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Gingival Overgrowth
Keywords: rotary; diode laser; gingivectomy; wound healing
MeSH Terms: conditions — Gingival Overgrowth | interventions — Lasers, Semiconductor; Laser Therapy

STUDY DESIGN:
Intervention Model Description: The trial is parallel-designed, controlled, prospective clinical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ceramic rotary bur (Experimental): For the ceramic bur group(Meisenger gingivectomies, ceramic rotary burs were used with 400-rpm rotary systems and with no serum irrigation, per the manufacturer's recommendation.
  Interventions: Device: Ceramic rotary bur
- Diode laser (Experimental): In the laser group (LG), a diode laser was applied to the operation sites in accordance with the manufacturer's guidelines (2.8 W continuous wave mode, wavelength 980 nm). The fiber optic laser tip had a 320-μm diameter with a 2.8 W output power. The laser never made contact with the gingival tissue. The practice distance did not affect the laser spot size, which was 0.5 cm-1 cm. Smoke associated with the laser application was aspirated from the surgical site.
  Interventions: Device: Diode laser
- Scalpel (Active Comparator): In the scalpel group following the local anesthetic administration, the gingivectomy was performed with a #15 scalpel. Subsequent to the operation, the borderline of gingiva was determined via the use of a pointer dental tweezers, and excessive gingival tissue was then removed with Gracey curettes
  Interventions: Device: Scalpel

INTERVENTIONS:
Device: Ceramic rotary bur — Gingivoplasties were performed with the same ceramic burs to easily provide a knife-edge appearance with ceramic rotary bur
  Other Names: Meisenger ceramic rotary bur
  Arms: Ceramic rotary bur
Device: Diode laser — The fiber optic laser tip had a 320-μm diameter with a 2.8 W output power were used in the study.
  Other Names: SiroLase Advance &Xtend
  Arms: Diode laser
Device: Scalpel — Scalpel surgery were performed as control group (conventioanl group).
  Arms: Scalpel

SUMMARY:
The aim of this study was to evaluate the degree of clinical discomfort and the issues experienced by patients and to use a software image program to compare wound healing during the 2-week period following gingivectomy performed with different techniques.

DETAILED DESCRIPTION:
Horizontal and vertical gingival overgrowth indexes were evaluated before and after surgery during each follow-up controls. The vertical distance of gingival tissue was measured from the gingival margin to the cement-enamel junction (gingival overgrowth [GO] index). Horizontal gingival values were also recorded between the tooth surfaces and the papillary tissue surface at the interdental contact point as buccolingual aspect (mesiobuccal [MB] index).

Postoperative Evaluations

The postoperative parameters, including pain, burning, edema, vascularization, erythema, epithelization, bleeding and carbonization, were recorded at 1, 3, 5, 7, and 14 days postoperatively.

Postoperative pain, burning, erythema, vascularization, and edema were assessed via the visual analogue scale (VAS). The VAS is a 100-mm horizontal-line scale that is used to quantify subjective symptoms such as pain, burning, erythema, vascularization, and edema. In the present study, researchers used a standard VAS on which patients drew a vertical sign along a 10-cm scale from 0 (no pain) to 10 (highest degree of pain). Bleeding and carbonization during the postoperative period were assessed as either present or absent. Patients evaluated their postoperative pain, burning, and bleeding values. The same researcher evaluated erythema, vascularization, edema, and epithelization values.

Evaluation of Surgical Wound Area After gingivectomy operation, the surgical site was evaluated with hydrogen peroxide to detect the presence of epithelization. A blinded researcher who used a standard digital camera to take standard magnification photographs assessed the operation area, consisting of the epithelium. The researcher examined all photographs with the assistance of an image-analyzing software program. The mesio-distal width of the maxillary right central tooth was recorded for each patient, and photographs were calibrated via the reference values. In the areas subjected to hydrogen peroxide application and experiencing tissue reaction, there was a lack of an epithelial layer in the wound area. The wound surface areas of foamy fields on the all of the groups' photographs were recorded on days 1, 3, 5, 7, and 14 following the gingivectomies.

ELIGIBILITY:
Inclusion Criteria:

The criteria for inclusion in the study were as follows:

* systemically healthy individuals
* nonsmokers
* horizontal and vertical gingival overgrowth indexes with a "score 1" or "score 2"
* mean bleeding on probing and mean plaque index value < 20% (indicating good oral hygiene)
* no clinical attachment loss and
* a minimum of four teeth at each surgical site.

Exclusion Criteria:

The exclusion criteria were as follows:

* systemic disease that could influence the outcome of the treatment, -pregnancy and/or lactation,
* allergy,
* conditions requiring antibiotic prophylaxis and anti-inflammatory medications, -acute or untreated periodontitis
* the use of an analgesic before the surgical procedure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Postoperative wound healing change | The wound surface areas of foamy fields on the all of the groups' photographs were recorded change between 1st day and 14th day following the gingivectomies.
  After gingivectomy operation, the surgical site was evaluated with hydrogen peroxide to detect the presence of epithelization

SECONDARY OUTCOMES:
Postoperative pain | Visual analogue Scale, minimum score is 0 and maximum score is 10.Change of VAS values were recorded on days between 1st and 14th days following the gingivectomies
  The Visual Analogue Scale is a 100-mm horizontal-line scale that is used to quantify subjective symptoms
Postoperative erythema | Visual analogue Scale, minimum score is 0 and maximum score is 10.Change of VAS values were recorded on days between 1st and 14th days following the gingivectomies
  The Visual Analogue Scale is a 100-mm horizontal-line scale that is used to quantify subjective symptoms
Postoperative burning | Visual analogue Scale, minimum score is 0 and maximum score is 10.Change of VAS values were recorded on days between 1st and 14th days following the gingivectomies
  The Visual Analogue Scale is a 100-mm horizontal-line scale that is used to quantify subjective symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ahu Uraz, PhD Dr, Study Director — Gazi University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giannelli M, Bani D, Tani A, Pini A, Margheri M, Zecchi-Orlandini S, Tonelli P, Formigli L. In vitro evaluation of the effects of low-intensity Nd:YAG laser irradiation on the inflammatory reaction elicited by bacterial lipopolysaccharide adherent to titanium dental implants. J Periodontol. 2009 Jun;80(6):977-84. doi: 10.1902/jop.2009.080648. PMID 19485829
- [Background] Tomasi C, Schander K, Dahlen G, Wennstrom JL. Short-term clinical and microbiologic effects of pocket debridement with an Er:YAG laser during periodontal maintenance. J Periodontol. 2006 Jan;77(1):111-8. doi: 10.1902/jop.2006.77.1.111. PMID 16579711
- [Background] Favia G, Tempesta A, Limongelli L, Suppressa P, Sabba C, Maiorano E. Diode laser treatment and clinical management of multiple oral lesions in patients with hereditary haemorrhagic telangiectasia. Br J Oral Maxillofac Surg. 2016 May;54(4):379-83. doi: 10.1016/j.bjoms.2015.08.260. Epub 2015 Sep 8. PMID 26360009